CLINICAL TRIAL: NCT04174781
Title: Preoperative Anti-PD-1 Antibody Plus Drug-eluting Bead TACE for BCLC Stage A/B Hepatocellular Carcinoma Beyond the Milan Criteria: A Phase II Trial
Brief Title: Anti-PD-1 Antibody Plus DEB-TACE for BCLC Stage A/B HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-5
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Immunotherapy

STUDY DESIGN:
Intervention Model Description: A Phase II Single-arm, Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEB-TACE+Sintilimab (Experimental): Participants with BCLC Stage A/B Hepatocellular Carcinoma Beyond the Milan Criteria
  Interventions: Drug: Sintilimab; Drug: DEB-TACE

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: 200mg iv Q3W D1
  Other Names: Immunotherapy; Anti-PD-1 therapy
Drug: DEB-TACE — DEB-TACE(epirubicin 60mg) D1; Additional DEB-TACE procedures were carried out every 4-6 weeks based on tumor response. A treatment cycle was defined as one DEB-TACE procedure plus two doses of sintilimab. The combination of DEB-TACE and sintilimab was continued for a maximum of 3 cycles until surgical resection, radiologic disease progression, unacceptable toxicity, or withdrawal from the study, whichever occurred first.
  Other Names: Drug-eluting Bead Transarterial Chemoembolization

SUMMARY:
This study aimed to evaluate the efficacy and the safety of the anti-programmed-death-1 antibody (anti-PD-1) Sintilimab Injection in combination with transarterial chemoembolization with drug-eluting beads(TACE-DEB) in patients with BCLC Stage A/B Hepatocellular Carcinoma Beyond the Milan Criteria.

DETAILED DESCRIPTION:
Patients with hepatocellular carcinoma (HCC) of BCLC stage A/B exceeding the Milan criteria have a low resection rate and high postoperative recurrence rate, therefore, optimizing therapy for these patients is an important unmet need. This study aimed to investigate the efficacy and safety of preoperative DEB-TACE plus sintilimab for the treatment of patients with BCLC stage A/B HCC exceeding the Milan criteria.

ELIGIBILITY:
Inclusion Criteria

1. Age between 18 years and 75 years;
2. ECOG PS 0/1;
3. Patients with histologically- or clinically-confirmed HCC (based on the American Association for the Study of Liver Diseases criteria) that was either BCLC stage A and exceeded the Milan criteria, or BCLC stage B
4. Have not received any anti-tumor systemic treatment in the past
5. No contraindications for the treatment of DEB-TACE and PD-1 inhibitors;
6. Liver function: Child-Pugh score Class A
7. The expected survival of the patient is more than 3 months
8. The following conditions must be met:

   Platelets ≥ 75 × 10^9/L White blood cell count (WBC) ≥ 3.0 × 10^9/L Hemoglobin ≥ 90 g/L Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN); total bilirubin (TBIL) ≤ 1.5 × ULN Blood creatinine ≤ 1.5 × ULN PT prolonged ≤ 3 s
9. Adequate bone marrow, cardiac, and renal function
10. Patients must agree to accept postoperative follow-up required by the design of this study;
11. Patients must have the ability to understand and voluntarily sign the informed consent, and must sign an informed consent before starting any specific procedure for the study.

Exclusion Criteria

1. History of other malignancies；
2. In combined with severe heart, lung, kidney or other important organ dysfunction, or combined with serious infection or other serious associated diseases, that cannot tolerate treatment (> CTCAE Version 5.0 adverse events of grade 2)；
3. With uncontrolled hepatitis B (HBV-DNA>2000 IU/ml and elevated ALT).
4. Spontaneous rupture and bleeding of HCC
5. Hepatic tumor burden >50% total liver volume
6. Complete occlusion of the portal vein
7. Evidence of a bleeding diathesis or coagulopathy, active infections, and autoimmune disease
8. Recurrent disease after surgery within the last 5 years
9. History of organ transplantation or plan to have liver transplantation;
10. Pregnant women, nursing mothers.
11. Patients have other factors that may interfere with patient enrollment and assessment results.
12. Refuse follow-up as required by this study protocol and refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per mRECIST | 36 months
  The duration from treatment initiation to PD in patients who cannot undergo surgery, or to the date of postoperative relapse in patients who receive surgery, or death for any reason, whichever occurs first (according to mRECIST).

SECONDARY OUTCOMES:
12 mo PFS rate | 36 months
  The percentage of patients who have not progressed or relapsed or death at the 12 mo time point since the first time of treatment.
Overall survival (OS) | 36 months
  The duration from treatment initiation to death from any cause.
Pathological Response | 6 months
  Including Major Pathological response rate（MPR）and pathological complete response (pCR). MPR is defined as the presence of 10% or fewer viable tumour cells in the primary tumours. pCR is defined as no viable tumour cells in the specimen.
Objective Response Rate (ORR) per mRECIST | 36 months
  The proportion of complete response or partial response as optimal response among all treated patients according to mRECIST.
Disease Control Rate (DCR) per mRECIST | 36 months
  The proportion of complete response, partial response or stable disease as optimal response among all treated patients according to mRECIST.
Adverse events (AEs) | 36 months
  The incidence, relationship with study drugs, and severity level of all adverse events (AEs) according to CTCAE 5.0, treatment-emergent adverse events (TEAEs), treatment related adverse events (TRAEs), and serious adverse events (SAEs) and the changes in vital signs, physical examination results, and laboratory test results before, during, and after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo C, Zhang J, Huang X, Chen Y, Sheng J, Huang X, Sun J, Xiao W, Sun K, Gao S, Que R, Shen Y, Zhang M, Wu J, Bai X, Liang T. Preoperative sintilimab plus transarterial chemoembolization for hepatocellular carcinoma exceeding the Milan criteria: A phase II trial. Hepatol Commun. 2023 Feb 9;7(3):e0054. doi: 10.1097/HC9.0000000000000054. eCollection 2023 Mar 1. PMID 36757445